CLINICAL TRIAL: NCT01426399
Title: A Randomized, Open-label, Multiple Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of LC15-0444 and Metformin After Oral Administration in Healthy Male Subjects
Brief Title: Pharmacokinetic/Pharmacodynamic Drug-drug Interaction of LC15-0444 and Metformin After Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DPCL009
Record Dates: First submitted 2011-08-22; First posted 2011-08-31 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; Metformin

ARMS (3):
- LC15-0444 (Experimental): LC15-0444 50mg qd
  Interventions: Drug: LC15-0444
- Metformin (Experimental): Metformin 1000mg bid
  Interventions: Drug: Metformin
- LC15-0444+Metformin (Experimental): LC15-0444 50mg qd +Metformin 1000mg bid
  Interventions: Drug: LC15-0444+Metformin

INTERVENTIONS:
Drug: LC15-0444 — LC15-0444 50mg qd (8 days once daily)
  Arms: LC15-0444
Drug: Metformin — Metformin 1000 mg bid (8 days twice daily)
  Arms: Metformin
Drug: LC15-0444+Metformin — LC15-0444 50mg qd (8 days once daily) + Metformin 1000 mg bid (8 days twice daily)
  Arms: LC15-0444+Metformin

SUMMARY:
The objective of the study was to investigate the drug-drug interaction between LC15-0444 and metformin by comparing the pharmacokinetic/pharmacodynamic, safety, tolerability in healthy male subjets after oral administration concomitantly and each alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 2months
* Subject who had whole blood donation in 2months, or component blood donation in 1months or transfusion in 1months currently.
* Smokers.(but, if the subject did'nt smoke in 3months, can participate the trial)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss | up to 171h30m
  To confirm and evaluate the pharmacokinetic characters of main metabolites of LC15-0444
Cmax,ss | up to 171h 30m
  To confirm and evaluate the pharmacokinetic characters of main metabolites of LC15-0444

SECONDARY OUTCOMES:
Vital signs | up to 171h30m
  to measure Safety and tolerability of the investigational products
AUECτ,ss | up to 171h30m
  Compare the pharmacodynamic interaction between LC15-0444 and metformin in healthy male subjects This parameter is been used to measure DPP4 activity
AUEC | up to 171h30m
  Compare the pharmacodynamic interaction between LC15-0444 and metformin in healthy male subjects This parameter is been used to measure Active/total GLP-1, glucose, insulin, c-peptide, glucagon.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D,Ph.D, Principal Investigator — Seoul national univ. hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin D, Cho YM, Lee S, Lim KS, Kim JA, Ahn JY, Cho JY, Lee H, Jang IJ, Yu KS. Pharmacokinetic and pharmacodynamic interaction between gemigliptin and metformin in healthy subjects. Clin Drug Investig. 2014 Jun;34(6):383-93. doi: 10.1007/s40261-014-0184-3. PMID 24627290